CLINICAL TRIAL: NCT03346902
Title: A Phase 2 Study to Evaluate Safety and Efficacy of EB-001 Injections in Facial Scar Reduction After Undergoing Mohs Surgery
Brief Title: Study of EB-001 in Facial Scar Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bonti, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB001-SR201
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Results first posted 2018-12-14 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Mohs Surgery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Drug: : Placebo: 0.9% Sodium Chloride Injection
  Injection of Placebo into area of scarring (forehead)
  Interventions: Drug: 0.9% Sodium Chloride Injection
- EB001 (Active Comparator): Drug: EB-001 Injection of EB-001 into area of scarring (forehead)
  Interventions: Drug: EB-001

INTERVENTIONS:
Drug: EB-001 — Injection of EB-001 into area of scarring (forehead)
  Arms: EB001
Drug: 0.9% Sodium Chloride Injection — Injection of Saline into area of scarring (forehead)
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of EB-001 in improving wound healing and reducing scar formation in patients undergoing Mohs surgery for skin lesions in the forehead area following a single treatment of EB-001 when injected into the muscles underlying the incision area.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of EB-001 in improving wound healing and reducing scar formation in patients undergoing Mohs surgery for skin lesions in the forehead area following a single treatment of EB-001 when injected into the muscles underlying the incision area.

The safety objective is to determine the safety and tolerability of single treatment of EB-001 when injected into facial muscles underlying a surgical wound during Mohs surgery.

The efficacy objective is to evaluate the efficacy of a single treatment of EB-001 when injected into the facial muscles (frontalis) underlying the surgical wound in improving wound healing, and reducing scar formation.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 75 years of age, inclusive
2. Subject in good health, or with stable treated medical condition, as determined by the investigator.
3. Scheduled to undergo Mohs surgery to remove a single skin lesion in the forehead. This could be

   1. Basal Cell Carcinoma
   2. Squamous Cell Carcinoma (non-metastatic)
   3. Other suitable lesions according to the investigator opinion
4. Lesion closure size at least 2 cm in length
5. Women of non-childbearing potential must be postmenopausal (at least 12 consecutive months of amenorrhea)
6. Women of childbearing potential must not be pregnant, lactating, or planning to become pregnant during the study
7. Women of childbearing potential agreeing to use either

   1. a highly effective method of contraception with failures rates less than 1% per year such as implant, intrauterine device (IUD), or sterilization from the day of dosing for 3 months (subjects who underwent sterilization must have initiated the procedure at least 3 months prior to the day of dosing) or
   2. dual methods of contraception with overall failures rates less than 1% per year such as injectable, pill, patch, ring, and diaphragm from the day of dosing for 3 months (subjects using oral contraception must have initiated treatment at least 2 months prior to the day of dosing)
8. Willing and able to complete and comply with procedures, protocol requirements and instructions, which includes completion of all required visits
9. Willing and able to sign and date IRB-approved informed consent
10. Able to speak, read, and understand the language of the informed consent form (ICF) and study questionnaires

Exclusion Criteria:

1. Pregnant or breast feeding, or planning a pregnancy
2. Body weight less than 50 kg (110 pounds)
3. Reported use of any botulinum toxin of any serotype within last 6 months before study drug administration
4. Anticipated use of any botulinum toxin of any serotype during the study
5. Known hypersensitivity to any botulinum toxin serotype
6. Known allergy or sensitivity to any of the components of the study treatments, or any materials used in the study procedures
7. Aminoglycoside intake within 48 hours prior to or during surgery
8. Pre-existing disorders of the neuromuscular junction (myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral Sclerosis)
9. Any uncontrolled medical condition that in opinion of investigator, puts subject at undue safety risk
10. Any clinically significant psychiatric condition that, in opinion of investigator, may interfere with study assessments or protocol compliance
11. Any cosmetic procedure, laser resurfacing treatment, or retinoid therapy in the forehead area in the past 30 days before study drug administration
12. Any eyebrow or eyelid ptosis at baseline as determined by the Investigator
13. History of hypertrophic scars or keloid formation or other wound abnormalities as assessed by the investigator
14. History of alcohol or drug abuse in the last 3 years, based on investigator judgement
15. User or former user of nicotine-containing products, as follows:

    1. including but not limited to cigarettes, cigars, and chewing or dipping tobacco) who stopped use or consumption (i.e., smoking, chewing, or pinching) of these nicotine-containing products less than 1 year before study drug administration, or
    2. topical or oral nicotine preparations for smoking cessation within the past 90 days before study drug administration
16. Anticipated need for surgery or overnight hospitalization during the study
17. Current enrollment in an investigational drug or device study or participation in such a study within 30 days or 5 half-lives of the drug, whichever is longer, of entry into this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earvin Liang, Study Director — Bonti, Inc.
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0.9% Sodium Chloride Injection: Single Injection of Saline into area of scarring (forehead)
- EB001: EB-001: Single Injection (0.5mL total) of EB-001 into area of scarring (forehead).
Period: Overall Study
Arm/Group | Placebo | EB001
Started | 4 | 8
Completed | 4 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EB001 | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Full Range); unit: years] | 67 [60 to 75] | 59 [34 to 72] | 62 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 8 | 12
Weight [Mean (Standard Deviation); unit: kg] | 87.28 (25.528) | 79.94 (19.352) | 82.38 (21.055)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Visual Analog Scale (VAS) Change (Values From 0 (Worst) to 10 (Best))
Description: Assessment of change in Visual Analog Scale score (values from 0 (worst) to 10 (best)) from day of surgery to Day 30. Percentage of subjects reporting an improvement in Visual Analog Scale score.
Time Frame: Day 30
Population: mITT
Measure: Number; unit: Percentage reporting improvement
Arm/Group | Placebo | EB001
Number analyzed (Participants) | 4 | 8
Percentage reporting improvement | 0 | 50

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Placebo | EB001
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | EB001 (N=8)
Asymmetry in facial features as a result of the temporal nerve being affected during the Mohs Surger (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03346902/Prot_SAP_000.pdf